CLINICAL TRIAL: NCT04147897
Title: Implementing mHealth for Schizophrenia in Community Mental Health Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dror Ben-Zeev, Professor, School of Medicine: Psychiatry And Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006141; 1R01MH116057-01A1 (NIH)
Record Dates: First submitted 2019-10-14; First posted 2019-11-01 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal Facilitation (Active Comparator): mHealth specialist is a trained clinician embedded in the clinical team offering the mHealth intervention, FOCUS.
  Interventions: Device: FOCUS
- External Facilitation (Active Comparator): mHealth specialist is a trained clinician external to the clinical team offering the mHealth intervention, FOCUS.
  Interventions: Device: FOCUS

INTERVENTIONS:
Device: FOCUS — FOCUS is a self management mHealth application for people with serious mental illness.

SUMMARY:
Randomized control trial examining two mHealth intervention strategies.

DETAILED DESCRIPTION:
The investigators will conduct a multi-site site hybrid type III effectiveness/implementation study in Washington State. The study involves a systematic head-to-head comparison between External Facilitation (EF) and Internal Facilitation (IF) implementation models applied to the FOCUS mHealth intervention.

ELIGIBILITY:
All participants need to be receiving clinical care at participating clinics who have partnered with the research team for this study.

Inclusion:

1. Chart diagnosis of SSD (i.e., schizophrenia, schizoaffective disorder, schizotypal disorder, delusional disorder, or schizophreniform disorder;
2. 18 years or older;
3. English-speaking;
4. Own a smartphone that can support FOCUS and active data plan.

Exclusion:

1. Used FOCUS in the past;
2. Plan to move or discontinue services at participating clinics in the upcoming 6 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dror Ben-Zeev, PhD, Principal Investigator — University of Washington
Locations (8):
- United States (8):
  - Cascade Mental Health Care, Chehalis, Washington
  - NEW Alliance Counseling Services, Colville, Washington
  - Compass Health, Everett, Washington
  - Valley Cities, Federal Way, Washington
  - Peninsula Behavioral Health, Port Angeles, Washington
  - Sound Health, Seattle, Washington
  - Frontier Behavioral Health, Spokane, Washington
  - Comprehensive Healthcare, Yakima, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Enrolled in study
Arm/Group | External Facilitation | Internal Facilitation
Started | 176 | 123
Completed baseline | 157 | 117
Completed | 157 | 117
Not Completed | 19 | 6
Period: 3M Follow up
Arm/Group | External Facilitation | Internal Facilitation
Started | 157 | 117
Completed | 101 | 85
Not Completed | 56 | 32
Period: 6M Follow Up
Arm/Group | External Facilitation | Internal Facilitation
Started | 101 | 85
Completed | 82 | 70
Not Completed | 19 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internal Facilitation | External Facilitation | Total
Number analyzed (Participants) | 117 | 157 | 274
Sex/Gender, Customized [Count of Participants; unit: Participants] — What best described you? Population: Analyzed includes only those that completed baseline assessment
  Participants
    Gender: Male | 64 | 75 | 139
    Gender: Female | 45 | 72 | 117
    Gender: Trandgender | 4 | 4 | 8
    Gender: Other | 4 | 4 | 8
    Gender: Unknown | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analyzed includes only those that completed baseline assessment
  Participants
    American Indian or Alaska Native | 3 | 9 | 12
    Asian | 3 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
    Black or African American | 12 | 17 | 29
    White | 81 | 108 | 189
    More than one race | 13 | 18 | 31
    Unknown or Not Reported | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analyzed includes only those that completed baseline assessment
  Participants
    Hispanic or Latino | 16 | 17 | 33
    Not Hispanic or Latino | 99 | 136 | 235
    Unknown or Not Reported | 2 | 4 | 6
Education [Count of Participants; unit: Participants] — What is the highest level of education you have completed? Population: Analyzed includes only those that completed baseline assessment
  Participants
    No formal school | 3 | 3 | 6
    Grade school | 1 | 2 | 3
    Junior high | 8 | 9 | 17
    High school diploma/GED | 72 | 109 | 181
    Associate's degree | 22 | 19 | 41
    Bachelor's degree or higher | 11 | 14 | 25
    Unknown | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Analyzed includes only those that completed baseline assessment
  Years | 43 (12) | 43.6 (11.7) | 43.4 (11.8)
Employment [Count of Participants; unit: Participants] — What is your current employment status? Population: Analyzed includes only those that completed baseline assessment
  Participants
    Unable to work / Disabled | 74 | 102 | 176
    Unemployed but looking for work | 14 | 13 | 27
    Unemployed but not looking for work | 2 | 7 | 9
    Employed full time | 6 | 11 | 17
    Employed part time | 14 | 12 | 26
    Student | 5 | 7 | 12
    Retired | 2 | 5 | 7
Housing [Count of Participants; unit: Participants] — What best describes your current housing status? Population: Analyzed includes only those that completed baseline assessment
  Participants
    Own/rent home or apartment | 78 | 99 | 177
    Friend's home or apartment | 23 | 31 | 54
    Mental health/substance use treatment facility or halfway house | 13 | 15 | 28
    Homeless | 2 | 11 | 13
    Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire (PHQ)-9
Description: The Patient Health Questionnaire (PHQ)-9 is the major depressive disorder (MDD) module of the full PHQ. Total scores range from 0-27. Higher scores represent more severe symptoms.
Time Frame: 0,3,6 months
Population: Baseline analyses include only those participants who completed baseline assessments (N=274; EF=157, IF=117). Participants who did not complete baseline assessments were excluded from analysis. 3M analyses include only those participants who completed 3M follow-up assessments (N= 186, EF=101, IF=85). 6M analyses include only those participants who completed 6M assessments (N=152, EF=82, IF=70).
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | External Facilitation | Internal Facilitation
Number analyzed (Participants) | 157 | 117
Scores on scale
  Baseline | 11.6 (0.5) | 10.7 (0.6)
  3M Follow-up: number analyzed (Participants) | 101 | 85
  3M Follow-up | 9.6 (0.6) | 10.2 (0.7)
  6M Follow-up: number analyzed (Participants) | 82 | 70
  6M Follow-up | 9.3 (0.7) | 9.4 (0.7)
Statistical Analysis 1: Comparison: External Facilitation vs Internal Facilitation; Mixed-effects linear models were used to analyze within-person changes from baseline to 3 months, accounting for repeated measures within participants and clustering of patients within agencies. Difference-in-differences estimates were derived to compare EF vs IF, with Cohen's d effect sizes calculated for each contrast; Test type: Superiority; p = .06, adjusted mixed-effects linear regression; Difference in Difference = 1.5; Cohen's d: 0.28
Statistical Analysis 2: Comparison: External Facilitation vs Internal Facilitation; Mixed-effects linear models were used to analyze within-person changes from baseline to 6 months, accounting for repeated measures within participants and clustering of patients within agencies. Difference-in-differences estimates were derived to compare EF vs IF, with Cohen's d effect sizes calculated for each contrast; Test type: Superiority; p = .25, Adjusted mixed-effects linear regression; Difference-in-Difference = 1.0; Cohen's d: 0.19

2. Primary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: The Generalized Anxiety Disorder-7 (GAD-7) measures generalized anxiety disorder symptoms. GAD-7 total score ranges from 0 to 21. Higher scores represent more severe symptoms.
Time Frame: 0,3,6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | External Facilitation | Internal Facilitation
Number analyzed (Participants) | 157 | 117
Scores on scale
  Baseline | 9.3 (0.5) | 9 (0.6)
  3M Follow-up: number analyzed (Participants) | 101 | 85
  3M Follow-up | 7.6 (0.6) | 7.9 (0.6)
  6M Follow-up: number analyzed (Participants) | 70 | 82
  6M Follow-up | 7.9 (0.7) | 7.6 (0.6)
Statistical Analysis 1: Comparison: External Facilitation vs Internal Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.37, adjusted mixed-effects linear regression; difference in difference = 0.7; Cohen's d: 0.13
Statistical Analysis 2: Comparison: External Facilitation vs Internal Facilitation; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .44, Adjusted mixed-effects linear regression; Difference-in-Difference = 0.6; Cohen's d: 0.13

3. Primary Outcome: Insomnia Severity Index (ISI)
Description: The Insomnia Severity Index (ISI) is a brief screening assessment tool designed to evaluate insomnia. Total scores range from 0-28. Higher scores represent more severe symptoms.
Time Frame: 0,3,6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | Internal Facilitation | External Facilitation
Number analyzed (Participants) | 117 | 157
Scores on scale
  Baseline | 12.4 (0.7) | 12.4 (0.6)
  3M Follow-up: number analyzed (Participants) | 85 | 101
  3M Follow-up | 11.4 (0.8) | 11.9 (0.7)
  6M Follow-up: number analyzed (Participants) | 70 | 82
  6M Follow-up | 12.6 (0.8) | 11.1 (0.7)
Statistical Analysis 1: Comparison: Internal Facilitation vs External Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .619, Adjusted mixed-effects linear regression; Difference-in-Difference = -0.4; Cohen's d: -0.07
Statistical Analysis 2: Comparison: Internal Facilitation vs External Facilitation; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.10, Adjusted mixed-effects linear regression; Difference-in-Difference = 1.5; Cohen's d: 0.26

4. Primary Outcome: Green Paranoid Thoughts Scale- Part B
Description: The Green Paranoid Thoughts Scale (GPTS)- part B measures ideas of persecution. Scores range from 16-80. Higher scores represent more severe symptoms.
Time Frame: 0,3,6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | Internal Facilitation | External Facilitation
Number analyzed (Participants) | 117 | 157
Scores on scale
  Baseline | 31.8 (1.7) | 32.5 (1.4)
  3M Follow-up: number analyzed (Participants) | 85 | 101
  3M Follow-up | 31.6 (1.8) | 30.4 (1.6)
  6M Follow-up: number analyzed (Participants) | 70 | 82
  6M Follow-up | 32.4 (1.9) | 30.1 (1.7)
Statistical Analysis 1: Comparison: Internal Facilitation vs External Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .32, Adjusted mixed-effects linear regression; Difference-in-Difference = 1.9; Cohen's d: 0.15
Statistical Analysis 2: Comparison: Internal Facilitation vs External Facilitation; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.16, Adjusted mixed-effects linear regression; Difference-in-Difference = 3.0; Cohen's d: 0.23

5. Primary Outcome: Symptom Check List (SCL-9)
Description: The Symptom Check List-9 (SCL-9) is a brief version of the SCL-90, which aims to evaluate a broad range of psychological problems and symptoms of psychopathology. Total scores are calculated as sum of all responses. Total sum scores range from 0-36. Higher scores mean more severe symptoms.
Time Frame: 0,3,6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | External Facilitation | Internal Facilitation
Number analyzed (Participants) | 157 | 117
Scores on scale
  Baseline | 13.7 (0.8) | 13 (0.9)
  3M Follow-up: number analyzed (Participants) | 101 | 85
  3M Follow-up | 11.2 (0.9) | 11.7 (1.0)
  6M Follow-up: number analyzed (Participants) | 82 | 70
  6M Follow-up | 10.7 (0.9) | 11.3 (1.0)
Statistical Analysis 1: Comparison: External Facilitation vs Internal Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .31, Adjusted mixed-effects linear regression; Difference-in-Difference = 1.1; Cohen's d: 0.15
Statistical Analysis 2: Comparison: External Facilitation vs Internal Facilitation; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .28, Adjusted mixed-effects linear regression; Difference-in-Difference = 1.3; Cohen's d: 0.17

6. Primary Outcome: Hamilton Program for Schizophrenia Voices Questionnaire (HPSVQ)
Description: A 9-item measure specifically designed to quantify characteristics of auditory hallucinations including frequency, negative content, loudness, duration, interference with life, distress, impact on self-appraisal, and compliance with commands. Total score is a sum of all 9 items. Total HPSVQ scores range from 0-36. Higher scores mean more severe symptoms.
Time Frame: 0,3,6 Months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | Internal Facilitation | External Facilitation
Number analyzed (Participants) | 117 | 157
Scores on scale
  Baseline | 14.3 (1.0) | 13.8 (0.9)
  3M Follow-up: number analyzed (Participants) | 85 | 101
  3M Follow-up | 13.6 (1.1) | 12.5 (1.0)
  6M Follow-up: number analyzed (Participants) | 70 | 82
  6M Follow-up | 13.0 (1.2) | 11.5 (1.0)
Statistical Analysis 1: Comparison: Internal Facilitation vs External Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .63, Adjusted mixed-effects linear regression; Difference-in-Difference = 0.5; Cohen's d: 0.07
Statistical Analysis 2: Comparison: Internal Facilitation vs External Facilitation; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .46, Adjusted mixed-effects linear regression; Difference-in-Difference = 0.9; Cohen's d: 0.12

7. Primary Outcome: Illness Management and Recovery Scales (IMRS)
Description: The Illness Management and Recovery Scales (IMRS) measure illness management and recovery. Scoring is a sum of all responses ranging from 15-75. Higher scores mean less severe symptoms.
Time Frame: 0,3,6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | External Facilitation | Internal Facilitation
Number analyzed (Participants) | 157 | 117
Scores on scale
  Baseline: number analyzed (Participants) | 101 | 85
  Baseline | 49.7 (0.7) | 49.8 (0.8)
  3M Follow-up: number analyzed (Participants) | 101 | 85
  3M Follow-up | 51.0 (0.8) | 50.7 (0.9)
  6M Follow-up: number analyzed (Participants) | 82 | 70
  6M Follow-up | 50.4 (0.8) | 51.2 (0.9)
Statistical Analysis 1: Comparison: External Facilitation vs Internal Facilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.67, Adjusted mixed-effects linear regression; Difference-in-Difference = -0.4; Cohen's d: -0.07
Statistical Analysis 2: Comparison: External Facilitation vs Internal Facilitation; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.53, Adjusted mixed-effects linear regression; Difference-in-Difference = 0.7; Cohen's d: 0.10

ADVERSE EVENTS:
Time Frame: Enrollment until end of follow-up, up to 24-weeks
Arm/Group | External Facilitation | Internal Facilitation
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/123
Other Adverse Events (participants affected / at risk) | 0/176 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT04147897/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT04147897/SAP_001.pdf
  • Informed Consent Form (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT04147897/ICF_002.pdf